CLINICAL TRIAL: NCT04744142
Title: Effects of Ketones on Muscle Wasting During Caloric Restriction in Lean Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Hespel, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S61133
Record Dates: First submitted 2021-01-25; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Muscle Wasting; Protein Intake; Ketosis; Caloric Restriction
Keywords: resting metabolic rate; β-hydroxybutyrate; caloric restriction; muscle mass; ketone ester
MeSH Terms: conditions — Muscular Atrophy; Ketosis

STUDY DESIGN:
Intervention Model Description: Subjects were pair-matched for body weight, % body fat and energy intake, where after they were randomly allocated to an experimental group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were randomized by an external, independent researcher. Supplements were color and taste matched.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (No Intervention): Received 10% protein in nutrition + placebo supplement
- Ketone (Experimental): Received 10% protein in nutrition + 3x20g B-hydroxybutyrate per day
  Interventions: Drug: Ketone supplementation
- High protein (Experimental): Received 30% protein in nutrition + placebo supplement
  Interventions: Dietary Supplement: Increased protein intake
- High protein + ketone (Experimental): Received 30% protein in nutrition + 3x20g B-hydroxybutyrate per day
  Interventions: Drug: Ketone supplementation; Dietary Supplement: Increased protein intake

INTERVENTIONS:
Drug: Ketone supplementation — Subjects receive either placebo or ketone ester supplementation
  Other Names: Placebo vs ketone supplementation
  Arms: High protein + ketone; Ketone
Dietary Supplement: Increased protein intake — Subjects receive either normal or increased protein intake
  Other Names: Normal vs increased protein intake
  Arms: High protein; High protein + ketone

SUMMARY:
Because of these anabolic properties of ketone bodies and the fact that ketone bodies prevent muscle protein breakdown for gluconeogenesis during energetic stress, ketone bodies can be a promising strategy to prevent or treat skeletal muscle wasting. Therefore, our aim is to investigate the effect of 3HHB intake on muscle wasting and its adverse consequences during a period of caloric restriction in lean females. In addition, we compare the effects of 3HHB intake with a high protein diet, which is currently considered as the best strategy to minimize lean loss during hypo-energetic periods. To end, we aim to investigate the synergistic effects of the intake of 3HHB in combination with a high protein diet.

DETAILED DESCRIPTION:
Thermodynamics state that body mass declines during periods in which energy expenditure exceeds energy intake. This negative energy balance can be obtained either by reducing energy intake, called caloric restriction, by increasing energy expenditure, i.e higher level of physical activity, or the combination of both. The sustained energy deficit results in a net loss of body weight due to losses of both fat and skeletal muscle mass in a ratio of approximately 3:11, depending on the severity of caloric restriction, diet composition and initial body fat percentage. Decreases in muscle mass are due to a combination of downregulated muscle protein synthesis in conjunction with an increased ubiquitin-proteasome-mediated muscle proteolysis, resulting in a negative net protein turnover.

In the context of sports, many athletes try to lose body weight to achieve different goals, such as improving performance by optimizing power-to-weight ratio, competing in a certain body weight category or for aesthetic reasons. However, the loss of body weight is often accompanied by detrimental loss of skeletal muscle mass, which is associated with a myriad of negative consequences including impaired physical performance and increased susceptibility to injury. Hence, athletes undergoing periods of caloric restriction strive for body weight loss via fat loss, while minimizing loss of lean mass. Recent studies have demonstrated that an increased protein intake, higher than the recommended dietary allowance (0.8g/kg/day), attenuates the loss of muscle mass during caloric restriction. Research has shown that the high protein diet has minor effects on muscle proteolysis compared to normal dietary protein but restores muscle protein synthesis, which is probably the primary mechanism by which lean mass is preserved. Specifically, in young healthy athletes, it is shown that a higher protein intake of 1.6-2.4 g per kg body weight per day reduces the loss of muscle mass during short-term caloric restriction periods.

In female athletes, longer periods of low energy availability (with or without an eating disorder) are often interrelated with menstrual dysfunctions and decreased bone mineral density, a syndrome called the 'female athlete triad'. The triad is particularly common in sports that emphasize aesthetics or leanness and can impose lifelong health consequences. However, interventions that minimize loss of lean mass and prevent hormonal and bone metabolism dysregulations in females during periods of caloric restriction, are still missing.

Ketone bodies, i.e. D-β-hydroxybutyrate (βHB), acetoacetate (AcAc) and acetone are naturally occurring chemical compounds synthesized in the liver from circulating fatty acids under conditions of low blood glucose and insulin levels. In normal physiological conditions, the concentration of serum ketone levels remains low (< 0.1 mM). However, during starvation or applying a ketogenic diet, i.e low carbohydrate content, serum concentrations of βHB and AcAc can increase up to 5-8 mM and 1-2 mM, respectively. In these conditions, ketone bodies serve as an alternative and more efficient energy source for various tissues, including the brain, heart and skeletal muscle, thereby 'sparing' the glucose storages. In normal conditions, the brain can only use glucose as an energy fuel to maintain central nervous system functions. Therefore, sparing glucose storages during periods of energetic stress is extremely important for survival. Besides, this sparing of glucose storages prevents the breakdown of muscle proteins which can be used as precursors for gluconeogenesis, providing glucose for the brain and other tissues. Hence, the availability of ketone bodies reduces the breakdown of muscle proteins for gluconeogenesis and, thus, preserves skeletal muscle mass even when energy availability is limited. Therefore, elevating ketone body levels may be an important strategy to prevent skeletal muscle wasting during periods of energetic stress.

Since recently, serum levels of ketone bodies can be increased by the intake of the ketone body ester (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (3HHB). This orally absorbable ketone body ester is proven safe and well-tolerated in both animals and humans and can elevate ketone body levels within 30 min to 5-6 mM, similar to levels after approximately one week of fasting. The availability of this ketone body ester allows for controlled studies on the effect of ketone bodies on muscle homeostasis without the negative side-effects of starvation and a ketogenic diet, i.e high serum triglyceride and cholesterol levels. The effects of 3HHB on endurance performance is still debated. However, a recent study from our lab showed that post-exercise ingestion of 3HHB increases markers of protein synthesis, which was further confirmed by in vitro experiments. C2C12 myoblasts showed increased leucine-mediated muscle protein synthesis by incubation of physiological concentrations of ketone bodies. Most recently, we found that dietary supplementation with 3HHB substantially improved survival and maintenance of functional capacity and muscular integrity in a mouse model of cancer cachexia.

Because of these anabolic properties of ketone bodies and the fact that ketone bodies prevent muscle protein breakdown for gluconeogenesis during energetic stress, ketone bodies can be a promising strategy to prevent or treat skeletal muscle wasting. Therefore, our aim is to investigate the effect of 3HHB intake on muscle wasting and its adverse consequences during a period of caloric restriction in lean females. In addition, we compare the effects of 3HHB intake with a high protein diet, which is currently considered as the best strategy to minimize lean loss during hypo-energetic periods. To end, we aim to investigate the synergistic effects of the intake of 3HHB in combination with a high protein diet.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 40 years old
* Fat percentage between 16 and 25%
* Regularly involved in physical activity ( > 6 h/week)
* Use of hormonal contraceptives
* Good health status confirmed by a medical screening
* Stable body weight during the last 3 months prior to the study, i.e. no changes > 2 kg

Exclusion Criteria:

* Smoking
* Obsessive pursuit for thinness, evaluated by the Eating Disorder Inventory 3 (EDI-3) 'Pursuit of leanness' (i.e a score higher than 26/32) (see Appendix 5)
* Intake of any medication or nutritional supplement that is proven to affect exercise performance, except oral contraceptives
* Blood donation during the study
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 44 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Muscle mass | Muscle mass is measured before and after 4 weeks of caloric restriction
  The amount of muscle mass loss

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Koppo, PhD, Study Director — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
Results will be published in internationally peer-reviewed journals